CLINICAL TRIAL: NCT02467569
Title: Phase I Trial Evaluating Pharmacokinetics, Safety and Tolerability of the Irreversible Epidermal Growth Factor Receptor Inhibitor Hemay020 in Patients With Advanced Solid Cancer
Brief Title: Study Evaluating Hemay020 In Subjects With Advanced Solid Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Collaborators: Hainan General Sanyang Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hemay020P1 2014
Record Dates: First submitted 2015-06-02; First posted 2015-06-10 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Neoplasms，Non-Small Cell Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hemay020 (Experimental): Part one: Dose Escalation Group Hemay020 capsules will be taken orally in doses of 25mg, 50mg, 100mg, 200mg or 300mg once daily for 28 days.
  Part two: Extension Group Hemay020 capsules will be taken in two dose groups that assessed by Part one for 28 days.
  Interventions: Drug: Hemay020

INTERVENTIONS:
Drug: Hemay020

SUMMARY:
The purpose of this study is to assess the pharmacokinetics，safety and tolerability of Hemay020 and to determine the recommended dose for future Phase II study as well as to obtain preliminary information on the efficacy of Hemay020 in subjects with solid tumors. The study will be conducted in two parts. Part one, testing will be done on up to 16-31 subjects to determine the safety and tolerability of Hemay 020 in patients with advanced solid tumors. Part two, another 16-24 subjects with advanced or metastatic NSCLC, will be added to the trial to better define the tolerability and preliminary efficacy of Hemay020.

DETAILED DESCRIPTION:
This is a phaseⅠsequential-group study of ascending single and multiple oral doses administered to subjects with advanced solid tumors. Each subject will receive a single dose of Hemay020, followed by a 2-week observation period, and then will receive Hemay020 administered once daily by mouth for 28 days. Each cycle consist of 28 days. Subjects will be enrolled in groups of 3 to 6. Depending on the safety and activity profile observed during the dose escalation phase, the dose selected for Part 2 may be adjusted. Part 2 is an extension part of two dose groups administered to subjects with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 70 years;
2. Subjects with histologically or cytologically confirmed diagnosis of solid tumor; and subjects who have failed standard therapy，or no effective therapy available for such patients;
3. at least one measurable tumour lesion (non radiation field) as defined by RECIST criteria and measured by CT or MRI techniques;
4. Patients have received chemotherapy at least 4 weeks prior to screening and must have recovered from any toxic effects of the treatment to CTCAE≤Grade 1;
5. Part 1 Only: ECOG Performance Status of 0,1;
6. Life expectancy of at least three (3) months;
7. Adequate bone marrow, liver, kidney and coagulation function, meeting the following criteria:

   ANC≥1.5×109/L，HB≥90g/L，PLT≥75×109/L； TBIL≤2×ULN； ALT≤2.5×ULN，AST≤2.5×ULN（ALT≤5×ULN，AST≤5×ULN if liver metastases are present） Serum creatinine≤1.5×ULN INR≤1.5×ULN Patients without gastrointestinal tract disease, which results in malabsorption syndrome, or patients who are unable to take oral medication;
8. All female and male subjects must agree and commit to the use of two contraceptive regimen for the duration of the study and for 6 months after the last dose of test article. Female subjects must have a negative serum or urine pregnancy test performed within 72 hours prior to treatment. Male subjects's sexual partner must use two contraceptive regimen.

   Two contraceptive regimens include a medication and non-medication contraceptive regimen;
9. Able to understand and sign a written informed consent before study entry;

   Inclusion Criteria for Part 2 Only:
10. Histological or cytological diagnosis of EGFR wild-type (or genetype is not determined) patients, with advanced or metastatic lung cancer after receiving two chemotherapy; or advanced or metastatic patients with EGFR mutation after receiving EGFR-TKI and one chemotherapy.
11. ECOG Performance Status of 0,1,2

Exclusion Criteria：

1. Patients with parenteral nutrition; malabsorption syndrome; any condition possibly affecting drug absorption or inability to tolerate oral medications;
2. Immunodeficiency history, including human immunodeficiency HIV positive（by ELISA and Western Blot）;
3. clinically QTc prolongation, ventricular tachycardia, ventricular fibrillation, heart block, myocardial infarction within 1 year, congestive heart failure, symptoms requiring medicine treatment patients with coronary heart disease;
4. Left ventricular ejection fraction (LVEF) <40％;
5. active infection (ie, requiring intravenous antibiotic or antiviral agent);
6. Organ or system status:

   * Patients with brain metastasis untreated surgical resection or radiotherapy, Patients with treated brain metastasis may be excluded if they are neurologically unstable and have been on steroids or receiving steroids less than 4 weeks prior to study;
   * Patients with bone marrow metastasis;
   * Documented history of interstitial lung disease, drug induced interstitial lung disease, radiation pneumonitis with steroids treatment, any evidence of clinically active interstitial lung disease;
   * Idiopathic fibrosis of the lung by CT scan before study entry;
   * Presence of clinically significant or uncontrolled disease (ie. unstable or uncompensated respiratory, heart, liver, kidney disease) in the investigator's judgment;
   * Any unstable systemic disease(including severe hypertension, unstable angina, congestive heart failure, liver and kidney or metabolic disease)
   * Any other malignant cancer within 5 years with the exception of adequately treated cervical cancer in situ or basal and squamous cutaneous cell carcinomas
   * Neurological and psychogenic disorders, including epilepsia or dementia;
7. Major surgery (not including biopsy) or injury within 4 weeks of treatment day 1;
8. History of alcohol or drug abuse;
9. Women who are pregnant or breast feeding or plan to be pregnant;
10. Pulse rate<40 per minute or >120 per minute; systolic pressure>140mmHg or diastolic pressure>90mmHg; axillaty temperature ≥37.1℃ or oral temperature ≥37.3℃;
11. Have a known hypersensitivity to the test article or any of the excipient of the test article;
12. Have received other clinical trials treatment within the last 3 months or at the time of study;
13. History of herbal ingredient, depressant, hypnotic or other drug abuse;
14. Evidence of significant medical illness or abnormal laboratory finding that would make the subject inappropriate for this study in by the investigator's judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07-03 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | At screening, weekly up to 18 months
Observed maximum concentration of Hemay020 | 0, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 hours post-dose on day 1 and day 42
Time of maximum concentration of Hemay020 | 0, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 hours post-dose on day 1 and day 42
Area under the plasma concentration versus time curve of Hemay020 | 0, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 hours post-dose on day 1 and day 42
Trough Plasma Concentrations of Hemay020 | 0, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144 hours post-dose on day 1 and day 42
Predose plasma concentration | Predose on day 8, 15, 22]

SECONDARY OUTCOMES:
Disease control rate (complete response rate + partial response rate + stable disease rate) according to RECIST v1.1 | At screening, after 4 weeks of treatment
Objective response rate (complete response rate + partial response rate) according to RECIST v1.1 | At screening, after 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Haiying Wu, Professor, Principal Investigator — Sun Yat-sen University Cancer Centre
Locations (1):
- Sun Yat-Sen University Cancer Centre, Guangzhou, Guangdong, China